CLINICAL TRIAL: NCT05151081
Title: The Role of Primary Nocturnal Enuresis in the Etiology of Overactive Bladder Syndrome
Brief Title: Overactive Bladder Syndrome
Status: Completed | Type: Observational
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Other Study IDs: 2020/04
Record Dates: First submitted 2021-11-11; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Overactive Bladder Syndrome; Enuresis, Nocturnal
Keywords: Overactive bladder; Enuresis nocturna; treatment; etiology
MeSH Terms: conditions — Nocturnal Enuresis; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Enuresis, Non-Enuresis: Patients were divided into two gruops according to whether having NE or not during childhood
  Interventions: Other: basicly

INTERVENTIONS:
Other: basicly — Do not repeat information already included in arm/group descriptions.

SUMMARY:
Purpose:

A lot of etiological factors related to overactive bladder (OAB) has been investigated. However, the role of primary nocturnal enuresis (NE), which is characterized with childhood night time incontinence, in the etiology of OAB is controversial. This study aims to evaluate the effect of NE in patients diagnosed with OAB.

Metod Between january-september 2021, the data of patients who applied to the urology outpatientclinic with OAB symptoms were collected. Patients with a history of chronic systemic disease, previous medical treatment for OAB and who did not accept to join the study were excluded. According to the diagnosis of childhood NE, patients were divided into two groups. Demographic data hav been recorded. Frequency of incontinence, number of day time void and nocturia were evaluated according to a 3 day voiding diary. Inaddition, max. Urinary flowr atio (Qmax), bladder Wall thickness and postvoid residual volüme rates were determined using uroflowmetry and pelvic ultrasound.

DETAILED DESCRIPTION:
A prospective randomized study is a study based on basic urological data. This study aims to evaluate the effect of NE in patients diagnosed with OAB.

ELIGIBILITY:
Inclusion Criteria:

* overactive bladder syndrome
* enuresis nocturna

Exclusion Criteria:

* diabetes mellitus,
* neurological diseases
* bladder outlet obstruction,
* active urinary system infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: up to 18 year and all sex
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
A diagnose of childhood NE in OAB patients can cause more severe semptomatologic progression | 1 years
  This study aims to evaluate the effect of NE in patients diagnosed with OAB.Definition of NE is urinary incontinence in children over the age of 5 during sleep ,as defined by International Children's Continence Society.
  Overactive Bladder Symptom Score (OABSS) questionnaire were used for the assessment of OAB. OABSS is an questionnaire ,consisting of 4 questions, was prepared by Homma et al. in 2006

CONTACTS AND LOCATIONS:
Overall Officials: Basri Cakiroglu, Study Chair — Hisar Intercontinental Hospital
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No